CLINICAL TRIAL: NCT04593823
Title: A Multicenter, Randomized, Open Label, Controlled Study Evaluating the Effectiveness and Safety of Furoscix On-Body Infusor vs Continued Medical Therapy for Worsening Heart Failure
Brief Title: Avoiding Treatment in the Hospital With Furoscix for the Management of Congestion in Heart Failure - A Pilot Study
Acronym: AT HOME-HF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: scPharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: scP-01-008
Record Dates: First submitted 2020-10-02; First posted 2020-10-20 (Actual); Results first posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Furoscix Infusor (Experimental): Furoscix (furosemide injection, 8 mg/mL) administered subcutaneously over 5 hours via the Furoscix Infusor. The Infusor is applied to the abdomen via a medical grade adhesive and delivers a subcutaneous infusion of Furoscix through a pre-programmed, biphasic delivery profile with 30 mg (3.75 mL) administered over the first hour, followed by 12.5 mg (1.56 mL) per hour for the subsequent 4 hours (Total dose is 80 mg (10 mL) over 5 hours).
  Interventions: Combination Product: Furoscix Infusor
- Continued Medical Therapy (No Intervention): The subjects enrolled in this arm will receive treatment as usual

INTERVENTIONS:
Combination Product: Furoscix Infusor — Furoscix Infusor, a drug-device combination product for subcutaneous delivery of Furoscix, buffered furosemide injection, 8 mg/mL (total dose = 80 mg dose) administered subcutaneously for 5 hours.
  Arms: Furoscix Infusor

SUMMARY:
This is a multicenter, randomized, open label, controlled study evaluating the effectiveness, and safety of the Furoscix Infusor vs continued medical therapy in patients with chronic heart failure and fluid overload requiring augmentation in diuretic therapy outside of acute care setting.

The study drug, Furoscix (furosemide injection 8 mg/ml), is a furosemide solution buffered to a neutral pH containing 80 mg/10 mL for subcutaneous administration over 5 hours via the Furoscix Infusor.

The study objectives are:

1. To provide pilot data on the effectiveness and safety to inform a pivotal trial.
2. To inform population enrichment strategies
3. To refine pivotal trial endpoints and analytical methods
4. To identify operational challenges of study design
5. To assess patient adherence, competence, and experience
6. To familiarize staff and patients with device application and use

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness and safety of the Furoscix Infusor vs continued medical therapy in patients with chronic heart failure and fluid overload requiring augmentation in diuretic therapy outside of acute care setting. 51 patients will be randomly assigned (2:1) to receive Furoscix vs continued medical therapy.

The Treatment Phase comprises a pre-programmed bi-phasic 5-hour drug administration of Furoscix (80 mg/10 mL) via the On-body Infusor. Subjects and/or their caregivers will be trained on device preparation, placement and removal in accordance with product instructions of use (IFU). Subjects should be transitioned back to their oral maintenance diuretic regimen when clinically indicated at the discretion of the investigator.

Over the initial 7 days, all subjects will receive daily clinic or phone follow-up by the study staff. Decision of treatment with Furoscix in the intervention arm as well as changes in oral diuretic dosing in the control arm will be determined by the treating physician in coordination with the study nurse. Safety labs will be done on Days 1, 3, 7 and 30.

After Subjects have been transitioned to their oral maintenance diuretic regimen, additional doses of Furoscix (for Furoscix group) or IV diuretics (for Treat as Usual group) can be prescribed during the 30-day study period as needed based on the presence of congestion symptoms (e.g. dyspnea, edema, and/or excess weight gain) as determined by the investigator.

The Follow-Up Phase will include a visit to the clinic on Day 30 +/- 5 days where effectiveness and safety assessments will be performed including limited physical exam (including NYHA Class), Composite Congestion Score (CCS), 5-point Current Dyspnea Score, 7-point Dyspnea Score, vital signs, laboratory analyses, KCCQ-12, Visual Analog Score (VAS), 6MWT and adverse events.

ELIGIBILITY:
Inclusion Criteria:

Subjects are eligible for inclusion only if all the following criteria are met:

1. Age 18 years or older.
2. Diagnosis of symptomatic chronic heart failure (NYHA Class II-IV) with background loop diuretic therapy for at least 4 weeks.
3. Need for augmented diuresis outside of the acute care setting as determined by the investigator.
4. On background therapy including daily total furosemide equivalent dose (40-160 mg) of loop diuretic or equivalent.
5. The subject must have signs of volume expansion, defined as two or more of the following six signs:

   1. jugular venous distention
   2. edema (≥ 1+)
   3. ascites
   4. pulmonary congestion on chest x-ray
   5. pulmonary rales
   6. NT-proBNP ≥1000 pg/ml (1400 for patients in atrial fibrillation) or, for patients not on Entresto, BNP ≥200 (400 for patients in atrial fibrillation)
6. Increase over the preceding 30 days in at least one of the following symptoms characteristic of worsening heart failure:

   1. dyspnea
   2. fatigue
   3. exercise intolerance
7. Adequate environment for at home administration of Furoscix by patient or caregiver.

Exclusion Criteria:

A Subject is not eligible for inclusion if any of the following criteria apply:

1. Suspected high risk clinical instability with outpatient treatment.
2. Presence of a complicating condition, other than heart failure likely to require hospitalization in next 30 days.
3. Pregnant women or women of childbearing age who are not willing to use an adequate form of contraception.
4. Known allergy to the active and inactive ingredients of the study medication or device adhesive.
5. On experimental medication or currently participating in another interventional research study.
6. eGFR < 20
7. Serum potassium at baseline > 5.4 or < 3.6
8. Concomitant infection
9. Heart rate > 110
10. Received IV furosemide or bumetanide within last 24 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2021-05-03 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marvin A Konstam, MD, Principal Investigator — Principal Investigator; James E Udelson, MD, Principal Investigator — Principal Investigator
Locations (18):
- United States (18):
  - Heart Group of Eastern Shore, Fairhope, Alabama
  - The Heart Center Research, LLC, Huntsville, Alabama
  - Hartford Hospital, Hartford, Connecticut
  - Aventura Clinical Research, LLC, Aventura, Florida
  - University of Florida, Gainesville, Florida
  - Elite Cardiac Research, Hialeah, Florida
  - First Coast Cardiovascular Institute, Jacksonville, Florida
  - Cardiology Consultants, Pensacola, Florida
  - James A. Haley Veerans Hospital, Tampa, Florida
  - University Hospital - Augusta, Augusta, Georgia
  - Advocate Health and Hospitals, Downers Grove, Illinois
  - UnityPoint Health - Methodist Hospital, Peoria, Illinois
  - Michigan Heart, Ypsilanti, Michigan
  - St. Louis Heart and Vascular, St Louis, Missouri
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cone Health Medical Group, Greensboro, North Carolina
  - Lancaster General Hospital, Lancaster, Pennsylvania
  - University of Wisconsin, Madison, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Konstam MA, Massaro J, Dhingra R, Walsh M, Ordway L, Pursley MS, McLean DS, Saha S, Close N, Konstam JM, Luepke KH, Mohr JF, Udelson JE. Avoiding Treatment in Hospital With Subcutaneous Furosemide for Worsening Heart Failure: A Pilot Study (AT HOME-HF). JACC Heart Fail. 2024 Nov;12(11):1830-1841. doi: 10.1016/j.jchf.2024.07.015. Epub 2024 Sep 11. PMID 39269392

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 Screen Failures
Groups:
- Continued Medical Therapy: The subjects enrolled in this arm will receive Continued Medical Treatment as usual as per the investigator
Period: Overall Study
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Started | 34 | 17
Completed | 33 | 15
Not Completed | 1 | 2
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intention to Treat Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Furoscix Infusor | Continued Medical Therapy | Total
Number analyzed (Participants) | 34 | 17 | 51
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.5 (10.91) | 71.1 (11.03) | 66.0 (11.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 25 | 11 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 0 | 3
  Not Hispanic or Latino | 31 | 17 | 48
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 4 | 15
  White | 23 | 13 | 36
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Body Weight [Mean (Standard Deviation); unit: Kilograms (Kg)] | 112.56 (34.52) | 111.70 (30.7) | 112.28 (32.99)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 36.02 (7.88) | 36.59 (9.92) | 36.21 (8.52)
New York Heart Association Class [Count of Participants; unit: Participants] — Class I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, dyspnea.
  Class II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, dyspnea.
  Class III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  Class IV: Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest that worsen with physical activity.
  Participants
    Class I | 0 | 0 | 0
    Class II | 2 | 4 | 6
    Class III | 31 | 12 | 43
    Class IV | 1 | 1 | 2
NT-proBNP [Mean (Standard Deviation); unit: pg/mL] — N-terminal (NT)-pro hormone BNP (NT-proBNP) is a non-active prohormone that is released from the Heart in response to changes in pressure inside the heart.
  These changes can be related to heart failure and other cardiac problems. Population: 2 subjects missing NT pro-BNP from both groups
  pg/mL
    number analyzed (Participants) | 32 | 15 | 47
    (all) | 2249.4 (3208.04) | 5467.5 (4979.57) | 3276.4 (4096.51)
Daily Furosemide Equivalent Dose [Mean (Standard Deviation); unit: mg] — Loop diuretic doses were converted to furosemide equivalents with 1 mg bumetanide = 20 mg torsemide = 40 mg furosemide. Population: One subject was not receiving any oral loop diuretics at baseline
  mg
    number analyzed (Participants) | 33 | 17 | 50
    (all) | 146.7 (141.66) | 124.7 (115.01) | 139.2 (132.42)

OUTCOME MEASURES:

1. Primary Outcome: Win Ratio of Composite Endpoint
Description: Win Ratio calculated as number of pairs of Furoscix On-Body Infusor subject "wins" divided by number of pairs of Furoscix On-Body Infusor subject "losses" when compared to Continued Medical Therapy subjects.
  Components of Endpoint composite outcome: CV death, HF hospitalization, Urgent ED/Clinic visit at 30 days and percent change in NT-proBNP from baseline at Day 7.
  See Statistical Analysis Plan for detailed explanation of this statistical method.
Time Frame: Day 7, Day 30
Population: All randomized subjects
Measure: Number; unit: Number of Wins for the group
Groups:
- Continued Medical Therapy: The subjects enrolled in this arm received Continued Medical Treatment as usual as per the investigator
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Number of Wins for the group | 228 | 206
Statistical Analysis 1: Comparison: Furoscix Infusor vs Continued Medical Therapy; Test type: Superiority; Win Ratio = 1.11, 95% CI 2-sided [0.48 to 2.50] — A win ratio parameter signifies the percentage of wins that a treatment group has achieved when compared against a comparator

2. Primary Outcome: Number of Cardiovascular Deaths
Description: Total number of CV deaths between two groups
Time Frame: Baseline, 30 Days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Participants
  No | 33 | 17
  Yes | 1 | 0
Statistical Analysis 1: Comparison: Furoscix Infusor vs Continued Medical Therapy; Test type: Superiority; p > 0.999, Chi-squared; Mean Difference (Final Values) = 2.9, 95% CI 2-sided [-17.0 to 15.9]

3. Primary Outcome: Number of Heart Failure Hospitalizations
Description: Heart Failure hospitalizations compared between two groups
Time Frame: 30 Days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Participants
  No | 29 | 13
  Yes | 5 | 4
Statistical Analysis 1: Comparison: Furoscix Infusor vs Continued Medical Therapy; Test type: Superiority; p = 0.459, Chi-squared; Median Difference (Final Values) = -8.8, 95% CI 2-sided [-36.4 to 13.6]

4. Primary Outcome: Number of Urgent ED/Clinic Visits for Worsening Heart Failure
Description: Urgent ED/Clinic visits for worsening heart failure compared between two groups.
  Statistical analysis was not performed due to no ED/Clinic visits
Time Frame: 30 Days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Participants
  No | 34 | 17
  Yes | 0 | 0

5. Primary Outcome: NT-proBNP Change From Baseline
Description: Percentage change in NT-proBNP from baseline at Day 7 compared between two groups
Time Frame: 30 Days
Population: All randomized subjects
Measure: Median (Full Range); unit: percentage change from baseline (pg/mL)
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 30 | 11
percentage change from baseline (pg/mL) | -7.195 [-55.27 to 379.58] | -2.170 [-53.37 to 36.08]
Statistical Analysis 1: Comparison: Furoscix Infusor vs Continued Medical Therapy; Test type: Superiority; p = 0.547, ANOVA; Repeated measures analysis; Least Squares Mean Difference = 8.887, 95% CI 2-sided [-20.010 to 37.784]

6. Secondary Outcome: Number of Heart Failure Event Free Survival Days
Description: Out of 30 days, HF event-free survival is the average number of days subjects survived outside the hospital event-free.
Time Frame: 30 Days
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
days | 23.2 (4.79) | 14.3 (10.14)
Statistical Analysis 1: Comparison: Furoscix Infusor vs Continued Medical Therapy; Test type: Superiority; p = 0.336, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Number of Subjects Deceased or HF Event Occurred
Description: Subjects that are Deceased or HF event occurred (hospitalization for HF or urgent ED/clinic visits for HF) over 30 days compared between treatment groups.
Time Frame: 30 Days
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Participants
  No | 28 | 13
  Yes | 6 | 4

8. Secondary Outcome: Visual Analog Scale (VAS)
Description: The patient global assessment VAS is a patient-reported assessment of how good or bad a patient feels their health is on a given day. It is reported on a visual scale of 0 to 100, with 0 being the worst health they can imagine and 100 being the best health they can imagine.
Time Frame: Baseline, 7 Days, 30 Days
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
score on a scale
  Day 0 | 57.1 (18.12) | 48.8 (22.12)
  Day 7 | 66.8 (16.88) | 59.7 (23.27)
  Day 30 | 70.2 (18.47) | 60.7 (24.01)

9. Secondary Outcome: Composite Congestion Score (CCS)
Description: The composite congestion score (ccs) is calculated by summing the individual scores for orthopnea, pedal edema and jugular venous distension.
  The investigator-assessed the signs and symptoms of congestion (orthopnea, pedal edema, and jugular venous distension) on a 4-point grading scale ranging from 0 to 3.
  Higher score indicates greater severity of symptoms ranging from 0 to 9.
Time Frame: Baseline, Day 7, Day 30
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
score on a scale
  Day 0 | 3.9 (1.58) | 3.7 (1.72)
  Day 7 | 2.2 (2.18) | 2.6 (1.79)
  Day 30 | 1.5 (1.75) | 2.1 (2.52)

10. Secondary Outcome: 5-Point Current Dyspnea Score
Description: The 5-Point Current Dyspnea Status Questionnaire is a single-item, self-administered instrument that quantifies current symptoms of dyspnea. The scale includes the absence of dyspnea (a score of 1), mild shortness of breath (a score of 2), moderate shortness of breath (a score of 3), severe shortness of breath (a score of 4) and the worst possible shortness of breath (a score of 5)
Time Frame: Baseline, Day 7, Day 30
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
score on a scale
  Day 0 | 1.3 (1.0) | 1.8 (1.15)
  Day 7 | 0.8 (0.90) | 1.1 (0.93)
  Day 30 | 0.9 (0.82) | 1.3 (0.99)

11. Secondary Outcome: 7-Point Dyspnea Score
Description: The 7-Point Dyspnea Status Questionnaire is a single-item, self-administered instrument that quantifies changes in dyspnea symptoms since initiation of study product. The scale ranges from Markedly better, Moderately better, Minimaly better, No change, Minimally worse, Moderately worse to Markedly worse.
Time Frame: Baseline, Day 3, Day 7, Day 30
Population: All randomized subjects
Measure: Count of Participants; unit: Participants
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Participants
  Day 3: Markedly Better | 3 | 1
  Day 3: Moderately Better | 12 | 0
  Day 3: Minimally Better | 8 | 4
  Day 3: No Change | 8 | 8
  Day 3: Minimally Worse | 1 | 0
  Day 3: Moderately Worse | 0 | 1
  Day 3: Markedly Worse | 0 | 1
  Day 3: Missing | 2 | 2
  Day 7: Markedly Better | 4 | 2
  Day 7: Moderately Better | 13 | 3
  Day 7: Minimally Better | 5 | 4
  Day 7: No Change | 12 | 6
  Day 7: Minimally Worse | 0 | 0
  Day 7: Moderately Worse | 0 | 0
  Day 7: Markedly Worse | 0 | 0
  Day 7: Missing | 0 | 2
  Day 30: Markedly Better | 6 | 0
  Day 30: Moderately Better | 13 | 5
  Day 30: Minimally Better | 6 | 3
  Day 30: No Change | 5 | 6
  Day 30: Minimally Worse | 2 | 0
  Day 30: Moderately Worse | 1 | 0
  Day 30: Markedly Worse | 0 | 0
  Day 30: Missing | 1 | 3

12. Secondary Outcome: KCCQ-12 Summary Score
Description: The KCCQ-12 questionnaire is a patient-reported assessment to capture symptom frequency, physical and social limitations, and quality-of-life impairment as a result of HF, as well as an overall summary score. In the KCCQ-12, responses are given for each individual item is scored on a scale of 0-100 with higher scores indicating better health.
Time Frame: Baseline, 7 Days, 30 Days
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
units on a scale
  Baseline | 40.96 (18.296) | 30.54 (25.395)
  Day 7 | 51.55 (20.388) | 36.68 (24.074)
  Day 30 | 55.80 (24.480) | 45.33 (28.624)

13. Secondary Outcome: Six-Minute Walk Test (6MWT)
Description: Change from baseline in Six-Minute Walk Test (6MWT) across follow-up timepoints
Time Frame: Baseline, 7 Days, 30 Days
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
meters
  Baseline | 241.7 (115.89) | 177.6 (77.65)
  Day 7 | 269.0 (126.63) | 201.0 (85.32)
  Day 30 | 292.3 (112.76) | 192.3 (71.17)

14. Secondary Outcome: Percent Lung Fluid
Description: Lung fluid volume as measured via Remote Dielectric Sensing (ReDS)
Time Frame: Baseline, Day 7, Day 30
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: % Fluid Volume in Lungs
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
% Fluid Volume in Lungs
  Day 0 | 36.8 (6.41) | 34.5 (6.70)
  Day 7 | 34.8 (6.09) | 31.3 (6.25)
  Day 30 | 35.6 (6.60) | 34.4 (6.35)

15. Secondary Outcome: Body Weight
Description: Body weight of the patient on the day of visit
Time Frame: Baseline, Day 3, Day 7, Day 30
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: Kilograms
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
Kilograms
  Day 0 | 112.563 (34.516) | 111.704 (30.697)
  Day 3 | 110.748 (34.590) | 115.524 (30.942)
  Day 7 | 109.935 (33.996) | 116.199 (28.781)
  Day 30 | 110.357 (35.201) | 117.422 (30.879)

16. Secondary Outcome: Renal Function
Description: Change from baseline in serum creatinine
Time Frame: Baseline, Day 3, Day 7, Day 30
Population: All randomized subjects
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Furoscix Infusor | Continued Medical Therapy
Number analyzed (Participants) | 34 | 17
mg/dL
  Day 0 | 1.496 (0.608) | 1.696 (0.747)
  Day 3 | 1.611 (0.541) | 1.894 (0.861)
  Day 7 | 1.648 (0.747) | 1.811 (0.860)
  Day 30 | 1.641 (0.771) | 2.010 (1.147)

ADVERSE EVENTS:
Time Frame: 30 Days
Groups:
- Continued Medical Therapy: The subjects enrolled in this arm received treatment as usual as per the investigator.
Arm/Group | Furoscix Infusor | Continued Medical Therapy
All-Cause Mortality (participants affected / at risk) | 2/34 | 1/17
Serious Adverse Events (participants affected / at risk) | 12/34 | 4/17
Other Adverse Events (participants affected / at risk) | 23/34 | 9/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Furoscix Infusor (N=34) | Continued Medical Therapy (N=17)
Cardiac failure congestive (Cardiac disorders) | 7 | 4
Left ventricular hypertrophy (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1
Sudden cardiac death (General disorders) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Furoscix Infusor (N=34) | Continued Medical Therapy (N=17)
Cardiac failure congestive (Cardiac disorders) | 4 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 7 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Infusion site pain (General disorders) | 5 | 0
Infusion site bruising (General disorders) | 2 | 0
Asthenia (General disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 5 | 2
Nausea (Gastrointestinal disorders) | 3 | 0
Blood creatinine increased (Investigations) | 2 | 0
Pneumonia (Infections and infestations) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Dizziness (Nervous system disorders) | 0 | 1
Fatigue (General disorders) | 1 | 2
Weight increase (Investigations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-12-09): https://cdn.clinicaltrials.gov/large-docs/23/NCT04593823/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-07): https://cdn.clinicaltrials.gov/large-docs/23/NCT04593823/SAP_001.pdf